CLINICAL TRIAL: NCT06262880
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Investigate the Effects of a Dietary Supplement Containing N-trans-Caffeoyltyramine (NCT) and N-trans-Feruloyltyramine (NFT) on Gastrointestinal Barrier Function
Brief Title: Dietary Supplementation on Gastrointestinal Barrier Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brightseed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIO-2305
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Intestinal Permeability
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo treatment (Placebo Comparator): Placebo treatment (Microcrystaline cellulose): 1 capsule/d
  Interventions: Other: Microcrystaline cellulose (MCC)
- Active low dose of plant derived phenolics (Active Comparator): Active low dose of plant derived phenolics via 1 capsule/d
  Interventions: Dietary Supplement: plant derived phenolics
- Active high dose of plant derived phenolics (Active Comparator): Active high dose of plant derived phenolics via 1 capsule/d
  Interventions: Dietary Supplement: plant derived phenolics

INTERVENTIONS:
Dietary Supplement: plant derived phenolics — Dietary supplement containing plant derived phenolics
  Arms: Active high dose of plant derived phenolics; Active low dose of plant derived phenolics
Other: Microcrystaline cellulose (MCC) — Placebo treatment: Microcrystaline cellulose
  Arms: Placebo treatment

SUMMARY:
The purpose of the current study is to examine the effects of a dietary supplement containing plant derived phenolics at two different dose levels on parameters of gastrointestinal (GI) health in otherwise generally healthy adults with risk factors (high BMI and waist circumference) for increased GI permeability. The primary hypothesis is that supplementation with plant derived phenolics will improve gut health compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 30-69 years of age, inclusive at Visit 1 (Day -7).
2. BMI of ≥29.0 to <40.0 kg/m2 at Visit 1 (Day -7).
3. Waist circumference >102 cm for men and >88 cm for women.
4. Non-user or former user (cessation ≥12 months) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) with no plans to begin use during the study period.
5. Non-user of marijuana or hemp products within 6 months of Visit 1, with no plans to begin use during the study period. A washout of 7 days is required for topical products (e.g., lotions) and willing to refrain from use during the study.
6. Willing to maintain physical activity and exercise patterns, body weight, and habitual diet throughout the trial.
7. Willing to refrain from exclusionary medications, supplements, and products throughout the study.
8. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results.
9. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

1. Known sensitivity, intolerance, or allergy to any of the study products or their excipients.
2. Abnormal chemistry or hematology laboratory test result(s) of clinical significance at Visit 1 (Day -7), at the discretion of the Clinical Investigator. One re-test will be allowed on a separate day prior to Visit 2 (Day 0), for subjects with abnormal laboratory test results.
3. Clinically important diagnosed GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, gastroparesis / malabsorption conditions, eosinophilic disorders of the GI tract, and clinically significant lactose or gluten intolerance or other food allergies).
4. Recent (within 2 weeks of Visit 1; Day -7) history of an episode of acute GI illness such as nausea/vomiting or diarrhea (defined as ≥3 loose or liquid stools/d).
5. Self-reported history (within 6 weeks of Visit 1; Day -7) of constipation (defined as <3 bowel movements per week).
6. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (e.g., Parkinson's disease, multiple sclerosis, etc.), psychiatric (including depression and/or anxiety disorders) or biliary disorders. Conditions which are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
7. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at Visit 1 (Day -7). Stable use of hypertension medication is allowed [defined as no change in medication regimen within the 3 months prior to Visit 1 (Day -7)].
8. Received a COVID-19 vaccine within 2 weeks of Visit 1 (Day -7) or expect to receive a COVID-19 vaccine during the study period.
9. Received an influenza vaccine within 1 week of Visit 1 (Day -7). Influenza vaccine is allowed during the study but must not be received within 7 days prior to a study visit.
10. Had a positive SARS-CoV2 test and experienced symptoms for >2 months (i.e., "long-haulers").
11. Extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan/vegetarian) at the discretion of the Clinical Investigator.
12. History or presence of cancer (including any malignant GI polyps) within 2 years of Visit 1 (Day -7), except for non-melanoma skin cancer.
13. Major trauma or any other surgical event, including abdominal surgery which might influence GI function, within 3 months of Visit 1 (Day -7).
14. Signs or symptoms of an active infection of clinical relevance* within 5 days of Visit 1 (Day -7). The visit may be rescheduled such that all signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to Visit 1 (Day -7).
15. Antibiotic use within 1 month of Visit 1 (Day -7) and throughout the study period.
16. Regular use (i.e., >3 days/week) of anti-inflammatory medications (e.g., NSAIDS) within 1 month of Visit 1 (Day -7).
17. Use of medications (over-the-counter or prescription) and/or dietary supplements known to influence GI function, including but not limited to, pre- and probiotic supplements as well as foods or beverages containing live probiotics (e.g., yogurt, kombucha), fiber supplements, laxatives, enemas, suppositories, histamine H2 receptor antagonists, proton pump inhibitors, antacids, anti-diarrheal agents, and/or anti-spasmodic within 2 weeks of Visit 1 (Day -7) and throughout the study period. Standard multivitamin and mineral supplements are allowed.
18. Had a colonoscopy or endoscopy within 1 month prior to Visit 1 (Day -7).
19. Exposure to any non-registered drug product within 4 weeks prior to Visit 1 (Day -7).
20. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. Subjects who are pregnant during the study will be discontinued.
21. Female subjects who is unwilling to wear a tampon during the collection of the 24-h urine samples when these collections occur during the time of menstruation
22. Recent history (within 12 months of screening; Visit 1; Day -7) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
23. Has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

    * If an infection occurs during the study period, test visits will be rescheduled until signs and symptoms have resolved (at the discretion of the Clinical Investigator) at least 5 days prior to the scheduled study visits.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-02-06 (Estimated)

PRIMARY OUTCOMES:
0-2 h urine 13C Mannitol excretion | 0, and 42 days
  GI permeability will be assessed using a sugar probe (13C mannitol).

SECONDARY OUTCOMES:
2 to 8 h urine 13C Mannitol | 0, and 42 days
  GI permeability will be assessed using a sugar probe (13C mannitol).
0 to 2 h urine LMR | 0, and 42 days
  GI permeability will be assessed using a two-sugar (lactulose and 13C mannitol) probe procedure.
2 to 8 h urine LMR | 0, and 42 days
  GI permeability will be assessed using a two-sugar (lactulose and 13C mannitol) probe procedure. Two pooled urine samples (0-2 h and 2:01-8 h) will be collected over an 8 h period for subsequent analysis at Clinic.
Blood Biomarkers | 0, and 42 days
  Soluble CD14
Blood Biomarkers | 0, and 42 days
  LBP
Blood Biomarkers | 0, and 42 days
  I-FABP
Fecal Biomarkers | 0, and 42 days
  Secretory IgA
Fecal Biomarkers | 0, and 42 days
  Calprotectin
Inflammatory Biomarkers (Blood) | 0, and 42 days
  hsCRP
Inflammatory Biomarkers (Blood) | 0, and 42 days
  IL-1β
Inflammatory Biomarkers (Blood) | 0, and 42 days
  TNF-α
Inflammatory Biomarkers (Blood) | 0, and 42 days
  IL-6
7-day recall of gastrointestinal symptoms | 0, and 42 days
  Composite score of GITQ (sum of all 8 individual scores) Individual symptom GITQ score
7-day recall of gastrointestinal symptoms | 0, and 42 days
  Individual symptom GITQ score
Stool frequency | 0, and 42 days
  Bristol stool scale
Stool consistency | 0, and 42 days
  Bristol stool scale
Body Weight | 0, and 42 days
  Body Weight in kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Addison, Illinois, United States